CLINICAL TRIAL: NCT00362544
Title: Pilot Study on Safety of a Weekly Administration of 10mg/kg of AmBisome® in Antifungal Prophylaxis Treatment of Allogeneic Stem-cell Transplantation and Acute Leukaemia
Brief Title: PROPHYSOME: Pilot Study on Safety of a Weekly Administration of 10mg/kg of AmBisome® in Antifungal Prophylaxis Treatment of Allogeneic Stem-cell Transplantation and Acute Leukaemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GS-FR-131-104; GS-FR-131-0119
Record Dates: First submitted 2006-05-10; First posted 2006-08-10 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-07

CONDITIONS: Leukemia
Keywords: antifungal prophylaxis; allogeneic stem-cell transplantation; acute leukaemia; antifungal prophylaxis treatment of allogeneic stem-cell transplantation and acute leukaemia
MeSH Terms: conditions — Leukemia | interventions — liposomal amphotericin B

INTERVENTIONS:
Drug: Ambisome

SUMMARY:
This pilot study was designed in order to evaluate the safety and efficacy of an AmBisome loading dose regimen, in a weekly administration schedule, during the aplastic phase following induction or consolidation chemotherapy for acute leukaemia, and during the initial phase of allogeneic stem-cell transplant, which are both high risk periods as far as severe fungal infections development is concerned.

DETAILED DESCRIPTION:
This pilot study was designed in order to evaluate the safety and efficacy of an AmBisome loading dose regimen, in a weekly administration schedule, during the aplastic phase following induction or consolidation chemotherapy for acute leukaemia, and during the initial phase of allogeneic stem-cell transplant, which are both high risk periods as far as severe fungal infections development is concerned.

ELIGIBILITY:
Inclusion Criteria:

Male or female patients aged more than 18, Patients undergoing standard myelo-ablative, conditioning regimen and AGVHD ciclosporin prophylaxis for allogeneic stem cell transplantation, or Patients with acute leukaemia undergoing first induction therapy or second induction therapy after relapse, or consolidation therapy, Expected neutropenia < 0.5 giga/l for at least 2 weeks, Normal chest CT scan and/or normal X-ray of the chest at baseline, Patients with no sign or symptoms of fungal infection and no previous proven or probable IFI, Females of childbearing potential must be surgically incapable of pregnancy, or practising an acceptable method of birth control with a negative pregnancy test (blood or urine) at baseline, Understanding of the study and agreement of the patient to give written informed consent, Ability and agreement to comply with all study requirements, Patient willing to attend hospital appointments for each injection (infusions will be performed in hospital, under strict medical supervision). All patients will be hospitalised prior to, and remain in hospital for at least one day, after the first infusion.

Exclusion Criteria:

Known hypersensitivity to amphotericin B, in particular known history of anaphylactic reaction to amphotericin B, Patients undergoing cord transplantation, Creatinine clearance < 60 ml/min, Patient with moderate or severe liver disease as defined by AST or ALT > 5 times the upper limit of normal (ULN), Patients who are unlikely to survive more than 1 month, Febrile patients (≥ 38.5°C), Patients who have received systemic antifungal therapy within 15 days prior to the inclusion, Any severe cardiovascular disease (such as arrhythmias, in particular) which may constitute a contra-indication to AmBisome® administration, Any severe disease other than the haematological diseases described in the second inclusion criteria, which in the investigator's judgement may interfere with study evaluations or affect the patient's safety, Pregnant or nursing females, Patients previously included in this study, Patients who have taken any investigational drug in the last 30 days prior to the inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2003-10; Study Completion 2006-03

PRIMARY OUTCOMES:
The primary endpoint will be the safety defined by the incidence of adverse events occurring during the course of prophylaxis treatment (4 weeks for AL patients and 8 weeks for SCT patients).

SECONDARY OUTCOMES:
The secondary endpoints for assessing efficacy will be the following:
Incidence of probable or proven invasive fungal infection according to EORTC-MSG 35 criteria within the12 weeks following the initiation of prophylaxis treatment.
Incidence of fever of unknown origin requiring empirical antifungal treatment within 12 weeks after trial initiation.
Incidence of superficial fungal infections within 3 months after trial initiation.
Time differential for commencement of empirical antifungal treatment measured within 3 months after trial initiation.
Evidence of colonisation by fungal organisms observed within 3 months after trial initiation.
Survival rate at the end of treatment and incidence of mortality related to fungal infection within 12 weeks and 24 weeks after study drug initiation.
Renal toxicity
The incidence and grade of nephrotoxicity will be assessed.
Hepatotoxicity
The incidence and grade hepatotoxicity will be assessed.
Patients whose AST or ALT becomes > 10 times the ULN will be withdrawn from the study.
Ionic analysis
Hypokalaemia: its incidence and grade will be evaluated. Potassium supplements received by the patient will be recorded in the Case Report Form.
Hypomagnesaemia: its incidence and grade will be evaluated as well.
Laboratories used by both sites will provide a list of their reference ranges.
Ionic disorders should be corrected throughout the trial.
Cardiovascular toxicity
The most commonly reported cardiovascular adverse events are rhythm disorders. There is a risk of seeing their incidence increase if the infusion is given too quickly.
Vital signs and ECG will be monitored throughout the trial.
Patients will be withdrawn from the trial, if in the investigator's opinion, further participation may put them at risk.
General safety
All adverse events occurring during the trial will be reported in the CRFs.

CONTACTS AND LOCATIONS:
Overall Officials: Lamine Mahi, MD, Study Director — Gilead Sciences
Locations (1):
- Gilead Sciences, Paris, France